CLINICAL TRIAL: NCT03370159
Title: A Phase I/II Open-Label Dose Escalation Trial of CPI-613 in Combination With Docetaxel Chemotherapy as a Second-Line Treatment of Non-Small-Cell Lung Cancer
Brief Title: CPI-613 and Docetaxel in Treating Patients With Stage IIIB or IV Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decided not to move forward
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00044399; NCI-2017-02010 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 62217 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2017-12-04; First posted 2017-12-12 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Stage IIIB Non-Small Cell Lung Cancer AJCC v7; Stage IV Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — devimistat; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CPI-613, docetaxel) (Experimental): Patients receive CPI-613 IV over 2 hours on days 1 and 3, and docetaxel IV on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients that achieve stable disease after 6 courses then receive CPI-613 alone on days 1and 3. Courses repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 6,8-Bis(benzylthio)octanoic Acid; Drug: Docetaxel; Other: Pharmacological Study

INTERVENTIONS:
Drug: 6,8-Bis(benzylthio)octanoic Acid — Given IV
  Other Names: Alpha-Lipoic Acid Analogue CPI-613; CPI 613; CPI-613
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of 6,8-bis(benzylthio)octanoic acid (CPI-613) when given together with docetaxel and to see how well they work in treating patients with stage IIIB or IV non-small cell lung cancer. Drugs used in chemotherapy, such as CPI-613 and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerate dose (MTD) of CPI-613 when used in combination with docetaxel therapy in advanced stage non-small cell lung cancer (NSCLC). (Phase1) II. To evaluate the response rate in patients receiving CPI-613 in combination with docetaxel therapy. (Phase 2)

SECONDARY OBJECTIVES:

I. To determine the safety of CPI-613 addition to docetaxel therapy. II. To determine the progression-free survival with CPI-613 in combination with docetaxel therapy at 27 weeks.

III. To determine the median progression-free survival with CPI-613 in combination with docetaxel therapy.

OUTLINE: This is a phase I, dose-escalation study of CPI-613 followed by a phase II study.

Patients receive CPI-613 intravenously (IV) over 2 hours on days 1 and 3, and docetaxel IV on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients that achieve stable disease after 6 courses then receive CPI-613 alone on days 1and 3. Courses repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage IIIB or IV NSCLC with radiographic proof of measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
* Life expectancy of >= 3 months
* Patients must have received previous systemic therapy to include: a regimen of chemotherapy, immunotherapy including anti-PDL or anti-PD-L1 therapies, combined chemotherapy and immunotherapy, provided treatment was discontinued >= 2 weeks prior to initiation of treatment on the present protocol
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) within institutional upper limit of normal
* International normalized ratio (INR) =< 1.5 x upper limit of normal (ULN)
* Prothrombin time (PT) =< 1.5 x ULN
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN or within therapeutic range if receiving anticoagulant therapy OR
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study through 30 days after the last dose of study medication; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document (either directly or via a legally authorized representative)

Exclusion Criteria:

* Patients who have had immunotherapy or tyrosine kinase inhibitor (TKI) therapy within two weeks prior to entering the study
* Radiotherapy or prior systemic chemotherapy within 2 weeks
* Patients who have been treated with more than one chemotherapy regimen, immunotherapy regimen or chemotherapy/immunotherapy regimen for metastatic non-small cell lung cancer
* Adverse events resulting from previous therapies have not recovered to grade 1 or less
* Patients may not be receiving any other investigational agents
* Patients with untreated, symptomatic brain metastases should be excluded from this clinical trial (patients with asymptomatic brain metastases amenable to treatment with Gamma Knife radiosurgery ["GKRS"] are eligible and may receive GKRS while on protocol)
* Lactating females
* Patients with EGFR, ALK or ROS-1 mutations who are eligible for treatment with a TKI and who have not received such treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CPI-613 or docetaxel
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with CPI-613
* Any condition that may, in the opinion of the investigator, compromise the safety of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Phase II dose of 6,8-bis(benzylthio)octanoic acid (CPI-613) when administered in combination with a standard dose of docetaxel (Phase 1) | Up to 18 weeks
Response rate defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (Phase 2) | Up to 2 years
  Will estimate the proportion of patients with a response (complete response + partial response) and calculate a 95% confidence interval for this measure.

SECONDARY OUTCOMES:
Median progression-free survival (PFS) | From the start of treatment to the time of progression or death, assessed up to 2 years
  Will estimate the median PFS using standard survival methods (Kaplan Meier).
Number and degree of adverse events under the experimental therapy regimens graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | Up to 30 days after the last study drug is administered
  Will be estimated along with 95% confidence intervals for each adverse event. These estimates will be compared (not using specific statistical tests, but descriptively) to those reported in patients treated with docetaxel.
Overall survival (OS) | From the start of treatment to date of death, assessed up to 2 years
Progression-free survival (PFS) | From the start of treatment to the time of progression or death, assessed at 27 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Grant, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States